CLINICAL TRIAL: NCT03785587
Title: A Multi-Center Open-Label Extension Study to Assess the Long-Term Safety Tolerability and Pharmacokinetics of Sofpironium Bromide Gel 15% Applied Topically to Children and Adolescents Age 9-17 Years Previously Enrolled in BBI-4000-CL-105
Brief Title: A Safety Study of BBI-4000 Gel in Pediatric Patients With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI-4000-CL-108
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-12

CONDITIONS: Primary Axillary Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gel, 15% (Experimental): Sofpironium Bromide Gel, 15%, applied once daily to each axilla for 24 weeks
  Interventions: Drug: Sofpironium Bromide Gel, 15%

INTERVENTIONS:
Drug: Sofpironium Bromide Gel, 15% — Sofpironium Bromide Gel, 15%
  Other Names: BBI-4000

SUMMARY:
Hyperhidrosis is a disorder of abnormal excessive sweating. Primary hyperhidrosis (armpits, hands, and feet) affects approximately 4.8% of the US population and is believed to be caused by an overactive cholinergic response of the sweat glands. Sofpironium bromide (BBI-4000) is a novel soft-drug in development for the topical treatment of hyperhidrosis. This Phase 2 study will assess the long-term safety, tolerability, pharmacokinetics and efficacy of sofpironium bromide gel applied topically to pediatric subjects with axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is an open-label, phase 2 long-term study designed to evaluate the safety, local tolerability, pharmacokinetics and efficacy of sofpironium bromide gel when applied topically to the axillae.

Subjects will apply the gel once daily at bedtime, to both axillae.

A maximum of 24 subjects, will be enrolled to receive sofpironium bromide gel, 15%.

Adverse events, vital signs, and local tolerability assessments will be collected at each visit. Urine pregnancy tests will be taken throughout the course of the study for women of child bearing potential. Blood and urine samples will be collected and analyzed for pharmacokinetics, routine hematology, chemistry, and urinalysis parameters at specified visits. Patient-reported outcome assessments will be recorded during the study at predefined time points.

The study will be comprised of a total of 8 scheduled visits to take place over a 26 week period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥9 to <17 years of age in good general health.
* Diagnosis of primary axillary hyperhidrosis that meets all the following criteria: (a) HDSM-Ax of 2 - 4 inclusive at both the Screening Visit (Visit 1) and Baseline Visit (Visit 2). (b) Symptoms of axillary hyperhidrosis for greater than or equal to 6 months' duration prior to enrollment.

Exclusion Criteria:

* In the Investigator's opinion, any skin or subcutaneous tissue conditions of the axilla(e), (i.e., the axillary area should be deemed otherwise "normal", besides the hyperhidrosis diagnosis, and free of blisters, large boils or sinus tracts, significant scarring or open wounds).
* Prior use of any prohibited medication(s) or procedure(s) within the specified timeframe for the treatment of axillary hyperhidrosis: (a) Botulinum toxin to the axillary area within 9 months of enrollment. (b) Axillary thermolysis, sympathectomy or surgical procedures of the axillary area at any time in the past. (c) Serotonergic agonist (or drugs that increase serotonin activity including SSRIs), beta-blocker, alpha-adrenergic agonist (clonidine), dopamine partial agonist or tricyclic antidepressant treatment within 30 days of enrollment. However, if a subject has been on a stable dose (in the opinion of the PI) of any of these medications and has not had a recent change in hyperhidrosis frequency or severity for 3 months prior to enrollment; they may be included. Doses of these agents should not be altered during the course of the study. (d) Any topical treatment for hyperhidrosis, requiring a prescription, within 3 days of enrollment.
* Anticholinergic agents [with the exception of sofpironium bromide] used to treat conditions such as, but not limited to, hyperhidrosis, asthma, incontinence, gastrointestinal cramps, and muscular spasms by any route of administration (e.g., IV, oral, inhaled, topical) within 30 days of the enrollment.
* Use of potent oral inhibitors of cytochrome P450 CYP3A & CYP2D6 and transporter inhibitors (OCT2/MATE1/MATE2) 14 days prior to enrollment. The use of topical antifungal medications is permitted if not applied in the treatment area.
* Any oral or topical homeopathic or herbal treatment (i.e., alternative therapies such as sage tablets, chamomile, valerian root and St. John's Wort) within 14 days of enrollment.
* Use of any cholinergic drug (e.g., bethanechol) within 30 days of enrollment.
* Use of any anti-anxiety and/or anti-depressant, amphetamine product or drugs with known anticholinergic side effects is prohibited with the following exceptions: (a) If a subject has been on a stable dose of an anti-anxiety and/or anti-depressant drug and has not had a recent change in hyperhidrosis frequency or severity for 3 months; they may be included. (b) An amphetamine product may be allowed if the dose has been stable for greater than or equal to 6 months without change in hyperhidrosis frequency or severity for 3 months. (c) Drugs with known anticholinergic side effects (taken within the last 30 days), including dry mouth, blurred vision, may be allowed based on the Principal Investigator's assessment.
* Known causes of hyperhidrosis or known history of a condition that may cause hyperhidrosis (i.e., hyperhidrosis secondary to any known cause such hyperthyroidism, diabetes mellitus, medications, etc.).
* Subjects with hyperhidrosis symptoms initiated or exacerbated with menopause.
* Subjects with unstable type 1 or type 2 diabetes mellitus or thyroid disease, history of renal impairment, hepatic impairment, malignancy, glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, benign prostatic hyperplasia (BPH), neurological conditions, psychiatric conditions, Sjögren's syndrome, Sicca syndrome, or cardiac abnormalities that may alter normal sweat production or may be exacerbated by the use of anticholinergics in the Investigator's opinion.
* Known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Subject is pregnant, lactating or is planning to become pregnant during the study.
* Unable or unwilling to undergo multiple venipunctures.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD PhD, Study Director — Botanix Pharmaceuticals
Locations (1):
- Northwest Arkansas Clinical Trials Center, Rogers, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gel, 15%
Started | 21
Completed | 16
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Gel, 15%
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment Emergent Adverse Events (All TEAEs).
Description: Summarized by MedDRA LLT with a 3 point severity scale of mild, moderate and severe.
Time Frame: Through study completion (24 weeks).
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gel, 15%
Number analyzed (Participants) | 21
Participants
  Mild | 5
  Moderate | 5
  Severe | 0

2. Primary Outcome: The Number of Participants With Dermal Tolerability Symptoms of Burning, Stinging, Itching, Scaling or Erythema to the Axillae.
Description: Summary of local site tolerability by maximum severity symptom rating on a 5-point scale (0=absent, 1=minimal, 2=mild,-3=moderate, 4=severe)-Safety Population
Time Frame: Through study completion (24 weeks).
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Gel, 15% - MINIMAL ASSESSMENT; Gel, 15% - MILD ASSESSMENT; Gel, 15% - MODERATE ASSESSMENT; Gel, 15% - SEVERE ASSESSMENT: Sofpironium Bromide Gel, 15%, applied once daily to each axilla for 24 weeks
  Sofpironium Bromide Gel, 15%: Sofpironium Bromide Gel, 15%
Arm/Group | Gel, 15% - MINIMAL ASSESSMENT | Gel, 15% - MILD ASSESSMENT | Gel, 15% - MODERATE ASSESSMENT | Gel, 15% - SEVERE ASSESSMENT
Number analyzed (Participants) | 21 | 21 | 21 | 21
participants
  Burning | 1 | 1 | 2 | 0
  Stinging | 1 | 1 | 1 | 0
  Itching | 2 | 2 | 3 | 0
  Scaling | 1 | 0 | 0 | 0
  Erythema | 4 | 2 | 3 | 3

3. Primary Outcome: The Systemic Exposure (Ctrough) of Sofpironium and Its Primary Metabolite (BBI-4010)
Description: Trough levels of sofpironium based on sampling schedule.
Time Frame: Through study completion (24 weeks).
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Concentration Trough (ng/mL) Sofpironium Bromide Gel, 15%: Concentration Trough (ng/mL) Sofpironium PK Population N=20
- Concentration Trough (ng/mL) BBI-4010: Concentration Trough (ng/mL) BBI-4010 PK Population N=20
Arm/Group | Concentration Trough (ng/mL) Sofpironium Bromide Gel, 15% | Concentration Trough (ng/mL) BBI-4010
Number analyzed (Participants) | 20 | 20
ng/mL
  Week 0 | 0.12562 (0.326157) | 0.09364 (0.264432)
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 0.24386 (0.748205) | 0.08800 (0.203345)
  Week 24: number analyzed (Participants) | 16 | 16
  Week 24 | 0.04728 (0.173893) | 0.04438 (0.177500)

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Gel, 15%
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gel, 15% (N=21)
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dry Eye (Eye disorders) | 1
Mydriasis (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Chapped Lips (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Application Site Pain (General disorders) | 2
Application Site Pruritus (General disorders) | 2
Skin Infection (Infections and infestations) | 1
Decreased Appetitie (Metabolism and nutrition disorders) | 1
Burning Sensation (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied .

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT03785587/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT03785587/SAP_001.pdf